CLINICAL TRIAL: NCT01868698
Title: Effects of High Voltage Electrical Stimulation, Shortwave Diathermy and Kinesiotherapy on Arterial Blood Flow in the Lower Limbs of Diabetic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, PhD, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1143-8004
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes; Peripheral Arterial Disease
Keywords: Physical Therapy Modalities; Electric Stimulation Therapy; Hyperthermia, Induced; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Arterial Disease; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Kinesiotherapy (Experimental): Will be made active and resisted exercises of the lower limbs.
  Interventions: Other: Kinesiotherapy
- shortwave diathermy (Experimental): Will be applied for 20 minutes on the lower limbs.
  Interventions: Other: shortwave diathermy
- high-voltage electrical stimulation (Experimental): The therapeutic current will be applied for 20 minutes on lower limbs.
  Interventions: Other: high-voltage electrical stimulation

INTERVENTIONS:
Other: high-voltage electrical stimulation
  Arms: high-voltage electrical stimulation
Other: Kinesiotherapy
  Arms: Kinesiotherapy
Other: shortwave diathermy
  Arms: shortwave diathermy

SUMMARY:
Peripheral arterial disease (PAD) is a pathological condition limiting, resulting from a narrowing or occlusion of the artery diameter due to aneurysms, inflammation, atherosclerosis and thromboembolic events. One of the main risk factors for the development of DAP is diabetes mellitus due to its relation to the process of atherogenesis. Thus, the objective of this study is to evaluate the effects of three treatment modalities for PAD on the blood flow velocity. It is a crossover study. Fifteen women with diabetes receive three types of treatment, the order defined according draw: high voltage electrical stimulation, shortwave diathermy and kinesiotherapy. The blood flow of the lower limb will be assessed by Doppler ultrasound. The hypothesis of this study is that physical therapy resources increase the circulation of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Diagnosis of diabetes
* Diagnosis of peripheral arterial disease

Exclusion Criteria:

* Regular physical activity
* Smokers
* Thrombosis active
* Severe peripheral arterial disease

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Doppler ultrasound | 1 years
  Will evaluate the blood flow in the following arteries of the lower limbs: femoral, popliteal, posterior tibial and dorsalis pedis.

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Guirro, PhD, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.fmrp.usp.br